CLINICAL TRIAL: NCT00674492
Title: Patients' View of Hepatitis C Treatment Completion or Withdrawal
Brief Title: Hepatitis C Virus (HCV) Treatment Completion or Withdrawal
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SHP 08-193
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis C patients: patients who initiated antiviral treatment for hepatitis C

SUMMARY:
Qualitative pilot study of patients' views of their experience with antiviral treatment for hepatitis C.

DETAILED DESCRIPTION:
Qualitative pilot study of patient' views of their experiences with antiviral treatment for hepatitis C. Two groups of patients will be sampled: nine who completed a 24 or 48 week course of treatment and nine who withdrew from treatment prior to planned end. Interview data will be analyzed using narrative and grounded theory methods to identify attributes of treatment experience that may discriminate between completion and withdrawal.

ELIGIBILITY:
Inclusion Criteria:

Ever initiated anitiviral treatment for hepatitis C.

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VHA patients who ever initiated antiviral treatment for hepatitis C.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Clark, PhD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: patients who initiated antiviral treatment for hepatitis C
Period: Overall Study
Arm/Group | Group 1
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients who initiated antiviral treatment
Arm/Group | Group 1
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 57 [50 to 69]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Attributes of Treatment Experience
Description: Four basic reasons for persisting in antiviral treatment were identified: cure the disease, concern about diminishing time to act (avoid bad end), demonstation of personal strength, and redemption for past behavior.
Time Frame: Zero to five years since ending treatment.
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 21
participants
  Avoid Bad End | 14
  Perseverence | 15
  Achieve Cure | 7
  Redemption | 9

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes